CLINICAL TRIAL: NCT05379777
Title: Determination of Effective Dose 90 of Remimazolam That Can Maintain Loos of Consciousness From Sedation With Remimazolam in Adult Patients
Brief Title: Effective Dose of Remimazolam for Sedation in Patients Undergoing Lower Extremity Surgery Under Spinal Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Hajung Kim, Clinical Assistant Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1638
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Remimazolam; Orthopedic Procedures; Sedatives; Anesthesia, Spinal
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remimazolam (Experimental): A maintenance dose of remimazolam is administered for sedation
  Interventions: Drug: Remimazolam

INTERVENTIONS:
Drug: Remimazolam — Remimazolam The starting dose of remimazolam is 1 mg/kg/hr. If sedation does not proceed successfully, increase the infusion rate by 0.2 mg/kg/hr in the next patient. (However, if the infusion rate is less than 0.6mg/kg/hr, the dose is increased by 0.1mg/kg/hr.) If sedation has progressed successfully until the end of surgery, the next patient will use the same dose with a probability of 0.89 or 0.11 It is reduced by 0.2 mg/kg/hr with a probability of (However, if the infusion rate is 0.6mg/kg/hr or less, reduce it by 0.1mg/kg/hr.)

SUMMARY:
Currently used drugs for monitored general anesthesia include propofol, midazolam, and dexmedetomidine. Each drug has diﬀerent advantages and disadvantages. Remimazolam causes a relatively small decrease in blood pressure, and it has no injection pain. In addition, remimazolam has a very short onset time, and even after the continuous infusion, the onset of remimazolam is fast, and even after continuous injection, the eﬀect disappeared very quickly due to the short context-sensitive half time. and through continuous infusion, the patient's depth of anesthesia can be maintained constant. In addition, the short duration of action and the ability to quickly reverse the eﬀect of ﬂumazenil suggest that remimazolam can be used eﬀectively under general anesthesia as well as under general anesthesia. Remimazolam can be used as a continuous infusion for general anesthesia. However, it has also been reported to be used for sedation by continuous infusion or divided intravenous infusion. However, the eﬀective infusion dose of remimazolam for supervised general anesthesia without mechanical ventilation has not been established.

In this study, the ED90 of the maintenance dose that maintain loss of consciousness in patients when supervised general anesthesia is performed through continuous infusion of remimazolam after spinal anesthesia is obtained.

ELIGIBILITY:
Inclusion Criteria:

* ASA PS 1-3
* Patients undergoing lower extremity surgery under spinal anesthesia and sedation using remimazolam

Exclusion Criteria:

* Patients who refuse to participate in this study
* Patients with hypersensitivity to benzodiazepine or flumazenil
* Patients with severe renal/hepatic disease
* Patients with drug/alcohol abuse
* Patients who take antidepressants, anticonvulsants, psychoactive drugs chronically
* Patients with difficulty in communication
* Patients with severe obstructive sleep apnea or other airway problems
* Patients contraindicated to regional anesthesia
* Patients judged to be inappropriate for this study

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
success or failure of sedation maintenace | throughout the surgery
  MOAA/S score of 3 or less (MOAA/S: Modified Observer's Alertness/Sedation scale) Awake (5) - Unresponsive (0)

SECONDARY OUTCOMES:
Frequency of respiratory depression | throughout the surgery
  respiratory rate equal or less than 6 time per minute

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea